CLINICAL TRIAL: NCT03825549
Title: A Randomized Trial of Behavioral Economic Approaches to Reduce Unnecessary Opioid Prescribing
Acronym: REDUCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Donaghue Medical Research Foundation (Other); Sutter Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 829269
Record Dates: First submitted 2019-01-17; First posted 2019-01-31 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Acute Pain
Keywords: Opioids; Nudges; Emergency Medicine; Urgent Care; Feedback
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No intervention
- Individual Audit (Experimental): Clinicians will receive individual audit feedback informing them of their performance.
  Interventions: Behavioral: Individual audit feedback
- Peer Comparison (Experimental): Clinicians will receive peer comparison feedback informing them of how their performance compares to their peers.
  Interventions: Behavioral: Peer comparison feedback
- Individual Audit and Peer Comparison (Experimental): Clinicians will receive individual audit feedback informing them of their performance and peer comparison feedback informing them of how their performance compares to their peers.
  Interventions: Behavioral: Individual audit feedback; Behavioral: Peer comparison feedback

INTERVENTIONS:
Behavioral: Individual audit feedback — Practice sites randomly assigned to have individual audit feedback will be sent information by email to each clinician at the site each month for the duration of the intervention period. The email will inform the clinician that the health system is doing monthly audits and provide them the number of patients in the last month for whom they prescribed 30 opioid pills per prescription or higher.
  Arms: Individual Audit; Individual Audit and Peer Comparison
Behavioral: Peer comparison feedback — Practice sites randomly assigned to have peer comparison feedback will be sent information by email to each clinician at the site each month for the duration of the intervention period. Data on the mean number of opioid pills per prescription and the proportion of visits with an opioid prescription will be delivered using a 3-month rolling average as follows: a) If clinician is above median: informed how their data compares to the median; b) If clinician is below median but above 10th percentile: informed how their data compares to the 10th percentile; c) If clinician is 10th percentile or below: informed of their data and commended for being a "low prescriber."
  Arms: Individual Audit and Peer Comparison; Peer Comparison

SUMMARY:
In this study, the investigators will evaluate the effect of a health system initiative aiming to change clinician opioid prescribing behaviors using two behavioral economic interventions - individual audit feedback and peer comparison feedback of clinicians.

DETAILED DESCRIPTION:
Opioid-related abuse and overdose represent a growing national epidemic in the United States. Clinician practice patterns play an important role: opioid prescriptions impact the likelihood that patients will misuse or become dependent on these medications, with longer prescriptions leading to greater sustained use. In this study, we will evaluate a Sutter Health System quality improvement initiative using monthly individual audit feedback and/or monthly peer comparison feedback to clinicians to change opioid prescribing patterns. In partnership with Sutter Health System, this will be conducted using randomization to evaluate its effect. We will also conduct a process evaluation to understand factors associated with better or worse performance at the clinician level.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians

  1. Practiced primarily at participating emergency department or urgent care center
* Patients

  1. Presented to a participating emergency department or urgent care center during the study period
  2. Discharged to home from the visit

Exclusion Criteria:

* Clinicians

  1. Saw less than 100 patients in the prior year
  2. Practiced primarily at another site that is not in the main trial
  3. Did not practice at Sutter Health in the prior 90 days
* Patients

  1. Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Change in the mean number of pills per opioid prescription | Six months
  The primary outcome is the change in the mean number of pills prescribed per opioid prescription from baseline to the intervention period.

SECONDARY OUTCOMES:
Change in proportion of patient visits with an opioid prescription | Six months
  The secondary outcome is the change in proportion of patient visits in which an opioid is prescribed from baseline to the intervention period.

OTHER OUTCOMES:
Change in morphine milligram equivalents per opioid prescription | Six months
  The change in morphine milligram equivalents per opioid prescription from baseline to the intervention period.
Change in mean number of opioid pills per patient-visit | Six months
  The change in the mean number of opioid pills per patient-visit from baseline to the intervention period.
Change in proportion of patient-visits with non-opioid pain prescription | Six months
  The change in proportion of patient-visits with non-opioid pain prescriptions (e.g., ibuprofen, acetaminophen, celecoxib, or muscle relaxants such as cyclobenzaprine, baclofen or tizanidine) from baseline to the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania; Amol Navathe, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Sutter Heath, Walnut Creek, California, United States

IPD SHARING:
Plan to Share IPD: No